CLINICAL TRIAL: NCT00598416
Title: Psychoeducation for HCV and Alcohol Behaviors
Brief Title: Psychoeducation for Hepatitis and Alcohol Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NIAAA-NORTH-AA015201; R01AA015201 (NIH)
Record Dates: First submitted 2008-01-10; First posted 2008-01-21 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Hepatitis C; Substance Abuse
Keywords: Hepatitis C; Substance Abuse; Psychoeducation; Psychiatric functioning; Physical Functioning; Quality of Life; NIAAA; Alcohol
MeSH Terms: conditions — Hepatitis C; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Psychoeducation (Experimental)
  Interventions: Behavioral: Family-Responsive Psychoeducation Program (PERF)

INTERVENTIONS:
Behavioral: Family-Responsive Psychoeducation Program (PERF) — Group psychoeducation for HCV patients and their primary caregiver.

SUMMARY:
The proposed project will apply a unique, effective family-responsive psychoeducation program, PsychoEducation Responsive to Families (PERF), for Hepatitis C Virus (HCV) treatment. The goal is to demonstrate that the intervention will enlarge the eligibility of some patients for HCV treatment and help sustain others through it.

DETAILED DESCRIPTION:
This study aims to evaluate the utility of a psychosocial intervention (PsychoEducation Responsive to Families; PERF), applied to help patients prepare for and sustain HCV treatment in the treatment setting. Through careful psychiatric diagnosis and multiple longitudinal assessments, this study will also shed further light on the course of comorbid alcohol use, drug use, and other psychiatric syndromes and their interrelationships. The proposed study combines an innovative psychoeducation program with traditional HCV patient care and education. The goal of this work is to improve treatment adherence, allowing individual drug regimens to achieve their optimal effectiveness and reach a wider patient population. Support and sustenance of patients from a psychosocial perspective while they are in treatment should also help deliver more patients to sustained suppression of HCV as well as help presently untreated patients and populations become candidates for this therapy-ultimately reducing the disease burden of increasing numbers of patients needing liver transplantation or facing imminent death.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are seropositive for HCV as determined by ELISA test and confirmed by direct measure of viral load as part of their clinical care
2. Lack progressive or decompensated liver functions (manifest in jaundice, ascites, variceal bleeding, hepatic encephalopathy)
3. Age at least 18 years
4. Identified family member(s)/significant other(s) also willing to participate in the psychoeducation groups, and
5. Ability to provide informed consent for research participation. "Family" will be defined to include biological relatives, as well as any non-biological individual or significant other considered "family" by either the ill member or his/her immediate family.

Exclusion Criteria:

1. Inability to provide informed consent such as irreversible cognitive impairment precluding participation
2. Progressive or decompensated liver functions (manifest in jaundice, ascites, variceal bleeding, hepatic encephalopathy), and
3. Age <18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2006-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Increased treatment readiness and better treatment adherence for treatment of HCV. | Index, Post intervention, and 1 year follow-up

SECONDARY OUTCOMES:
Better management of substance abuse and other psychiatric disorders. | Index, Post intervention, and 1 year follow up
Better social functioning and increased quality of life. | Index, Post intervention, and 1 year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Carol S North, MD, MPE, Principal Investigator — Univeristy of Texas Southwestern Medical Center
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States